CLINICAL TRIAL: NCT05424198
Title: The Effectiveness and Procedural Characteristics of the Trident Multi-tined Cannula for Cervical Medial Branch Radiofrequency Ablation Compared to the Conventional Cannula; A Multi-site, Single Blinded, Randomized Controlled Trial
Brief Title: Trident Multi-tined Cannula for Cervical MBRFA Compared to the Conventional Cannula
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Allison Glinka Przybysz, Principle Investigator and Assistant Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB 143800
Record Dates: First submitted 2021-12-28; First posted 2022-06-21 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2024-06

CONDITIONS: Cervical Pain; Cervical Facet Joint Pain
Keywords: cervical medial branch radiofrequency ablation; cervical facet joint pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: To compare procedural characteristics, pain, and disability outcomes of cervical medial branch radiofrequency ablation (CMBRFA) using either a Trident or conventional cannula in patients with confirmed facet mediated pain (defined by ≥80% symptom reduction after dual medial branch block).
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be randomized to one of two standard of care procedures: trident cannula cervical medial branch radiofrequency ablation or conventional cervical medial branch radiofrequency ablation. Participants will be blinded to which group they are randomized to. Outcomes will be collected by a blinded third party.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Trident Cervical Medial Branch Radiofrequency Ablation (Active Comparator): During this procedure a 50 mm or 100 mm long (dependent on body habitus), 18-gauge insulated cannula with a 5 mm active tip will be placed perpendicularly at targeted medial branches (the nerves carrying pain signals from the facet joints).
  Interventions: Procedure: Cervical Medial Branch Radiofrequency Ablation
- Conventional Cervical Medial Branch Radiofrequency Ablation (Active Comparator): During this procedure a 50 mm or 100 mm long (dependent on body habitus), 18-gauge conventional cannula with a straight 5 mm active tip will be placed parallel and oblique to the targeted medial branch branches (the nerves carrying pain signals from the facet joints). At each location, one lesion will be made to accommodate anatomic variation.
  Interventions: Procedure: Cervical Medial Branch Radiofrequency Ablation

INTERVENTIONS:
Procedure: Cervical Medial Branch Radiofrequency Ablation — The skin and superficial tissues will be anesthetized at each site with 1-2 mL of lidocaine. Prior to the ablation up to 2 mL of lidocaine may be used at each site to ensure adequate pain control during the ablation. Once in position, a radiofrequency ablation lesion will be made using a 30 second ramp-up time to a maximum temperature of 80 °C, followed by an additional 90 seconds at maximum temperature.

SUMMARY:
Cervical medial branch radiofrequency ablation (CMBRFA) is an effective treatment for cervical facet pain. The efficacy of CMBRFA was proven by studies published in the late 1990's and early 2000's. Patients were selected by a strict, labor-intensive placebo-controlled, diagnostic block protocol and were treated using a conventional monopolar cannula that was positioned parallel to the medial branch, two to three lesions per medial branch nerve and both sagittal and oblique passes. Since the original CMBRFA publications, patient selection for CMBRFA is less strict, and new RFA cannulae have been developed to improve efficiency and safety while maintaining a large ablative lesion.

Current clinical patient selection criteria for CMBRFA tend to be more relaxed than described in early research studies. However, subsequent research has shown that when selection criteria are too relaxed, outcomes are poorer. A recent cross-sectional study reported that when CMBRFA is done in patients selected by >80% pain improvement after dual medial branch blocks, outcomes are similar to patients selected with a stricter selection protocol (100% pain relief) similar to the original CMBRFA studies. Although, the cross-sectional study suggests an appropriate selection criteria, it has not been used in any prospective studies.

The Trident multi-tined cannula is a recent technology that produces a large ablative lesion distal to the triple-tined tip. This design allows a perpendicular/lateral approach to CMBRFA and only requires a single lesion at each medial branch. This differs from the conventional cannula, which produces it's most extensive ablative lesion along the cannula with minimal distal projection. As a result, it requires a parallel approach with multiple burn cycles at the same medial branch. The perpendicular approach with Trident and single lesion cycle at each medial branch are appealing for safety purposes and efficiency however, it's efficacy has not been directly compared to the standard conventional cannula.

Problem: There are no randomized controlled trials comparing novel technologies like Trident cannula to the previously studied conventional cannula in patients selected with a more practical selection criteria.

Purpose: To compared procedural characteristics, pain, and disability outcomes of CMBRFA using either a Trident or conventional cannula in patients with confirmed facet mediated pain (defined by ≥80% symptom reduction after dual medial branch block).

Central Hypothesis: Trident cannula during CMBRFA will result in noninferior improvements in pain and function compared to conventional cannula but will significantly reduce procedural discomfort, time and radiation exposure.

Specific Aims:

1. Determine the proportion of patients with a successful pain response (defined as ≥50% improvement in index pain) to Trident (T-CMBRFA) versus conventional (C-CMBRFA) at 3, 6, and 12 months.
2. Determine the proportion of patients with a successful functional response (defined as ≥10% reduction on neck disability index [NDI]) to T-CMBRFA versus C-CMBRFA at 3, 6, and 12 months.
3. Determine the proportion of patients with a successful perception of improvement (defined as a score ≥6 on the Patient Global Impression of Change [PGIC]) to T-CMBRFA versus C-CMBRFA at 3, 6, and 12 months.

DETAILED DESCRIPTION:
According to the National Center for Health Statistics, neck pain is the third most commonly reported musculoskeletal complaint in the United States. Cervical zygapophysial or "facet" joint pain is responsible for at least 25% of patients with chronic neck pain and is higher in patients with neck pain after a whiplash injury. Individuals with verified facetogenic pain or cervicogenic headaches can be treated with cervical medial branch radiofrequency ablation (CMBRFA). CMBRFA is a minimally invasive percutaneous procedure that utilizes thermal energy to coagulate nerves from the facet joints, and thereby interrupt the nociceptive pain signals. The targeted nociceptive nerves are the medial branches of the cervical dorsal rami and the third occipital nerve.

The gold standard method of facet pain diagnosis is anesthetizing the medial branches that innervate the involved facet joint and subsequently evaluating the significance of symptom improvement; this process is known as a medial branch block (MBB). There is significant practice variability in what is considered a "positive" MBB. A single cervical MBB with 100% symptom improvement has a false positive rate of 27-60%. The false positive rate decreases with stricter selection criteria. The efficacy of CMBRFA was established in the late 1990's and early 2000's when using a strict selection criteria; 100% symptom improvement with concordant dual medial branch block ± placebo-control block.

In 1996, Lord et al. published in New England Journal of Medicine research showing that when the rigorous diagnostic criteria were adhered to, 63% (CI 95%: 57-69%) and 38% (CI 95%:32-44%) of patients were pain free at 6 and 12 months following CMFRFA. Though comparative dual MBB ± placebo with 100% symptom improvement reduces false positive rates, it is time consuming and expensive, exposes patients to extra radiation and procedural risk, is not required by insurance, and is not the Spine Interventional Society (SIS) recommended gold standard for patient selection for facetogenic pain in the lumbar spine. Currently insurance requires ≥80% symptom improvement with dual facet block. These insurance requirements are consistent with the research supported SIS guidelines for the diagnosis of lumbar facetogenic pain and such practical patient selection criteria are commonly utilized in clinical practice. A recent cross-sectional study reported that when CMBRFA is performed on patients selected by >80% symptom improvement after dual medial branch block, outcomes are similar to patients selected with a stricter selection protocol similar to the original CMBRFA studies however, this needs to be validated in prospective studies.

In early explanatory studies, providers used a conventional monopolar cannulae to ablate targeted medial branch nerves. C-CMBRFA cannula produce the largest lesions along the shaft of the cannula with minimal extension distal to the tip. To increase the likelihood of medial branch ablation the conventional cannula is placed parallel to the targeted medial branch in a posterior to anterior approach with sagittal and oblique passes, and 2-3 lesions per medial branch. Disadvantages to the conventional technique is the procedural time needed for multiple passes and burns and the risk of ventral advancement of the cannula towards vital neurovascular structures. Since the original explanatory C-CMBRFA studies, there have been technologic advances in RFA cannulae in an effort to improve safety and efficiency of CMBRFA.

The Trident multitined cannula was designed to allow a perpendicular/lateral approach to the medial branch nerves. Such approach results in point contact against bone, prevents unintended advancement towards neurovascular structures, and as a result adds to the safety of the procedure. There is also reported efficiency during Trident RFA since only 1 pass and a single lesion at each medial branch is required. A single burn cycle at each site is a possibility because of the unique lesion shape and size. The Trident cannula most commonly used for CMBRFA is 18-gauge and has a 5 mm exposed tip. Once the cannula tip is placed at the target location, 3 tines are deployed anterior and laterally from the cannula tip in an equilateral triangle configuration. Computer simulation calculations predict that a two-minute lesion at 75°C would result in thermal coagulation in an area measuring 7.6 mm wide by 7.6 mm length in the axial plane (at the periosteal surface) and 9.1 mm in height in the sagittal plane (soft tissue lesion) [data provided by Diros Technology Inc.]. These values are comparable to the findings of Finlayson et al who compared thermal lesions morphology of 2 multitined cannulae and a conventional monopolar cannula in an ex vivo model. In the axial plane, with the Trident cannula perpendicular to the periosteum, the mean lesion width and length were 7.3 x 8.8 mm respectively. In the sagittal plane, the mean lesion height was 7.3 mm. Considering that the mean distance between the medial branch nerve at the waist of the articular pillar, and the tip of the superior facet has been documented to be between 7.1-7.4 mm for C3 through C6 and 5.5 mm for C7, a single Trident lesion placed at the waist of the lateral mass should cover approximately one half of the periosteal surface. This should be adequate to accommodate medial branch nerve anatomical variation. Ultimately, the Trident cannula results in an approach that may be technically easier, quicker, safer, more comfortable and as effective as the traditional parallel/posterior approach however, there are no studies comparing Trident to conventional cannula during CMBRFA.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient aged ≥18 capable of understanding and providing consent in English and capable of complying with the outcome instruments used.
2. Axial (non-radicular) neck pain for at least 3 months.
3. 7-day average numeric pain rating score (NRS) for neck pain of 4/10 or greater at baseline evaluation.
4. *Positive responses to dual diagnostic MBB blocks using 0.5mL of lidocaine and bupivacaine, on respective encounters on separate days, at each of the appropriate MBBs.

   * Levels selected for diagnostic procedures will be determined by the treating physician based on the overall clinical picture including the location of pain, pain referral patterns, physical examination and imaging findings. The procedural techniques of all MBB blocks will be performed according to Spine Intervention Society guidelines.(14) A pain diary with appropriate diagnostic categories of relief will be provided (100% relief, 80-99% relief, etc.), will be provided. In order to qualify as a positive block, the subject must experience relief lasting at least one hour with lidocaine and two hours with bupivacaine.

Exclusion Criteria:

1. Those receiving remuneration for their pain treatment (e.g. disability, worker's compensation, auto injury in litigation or pending litigation).
2. The patient is incarcerated.
3. Those unable to read English and complete the assessment instruments.
4. Allergy to contrast media or local anesthetics.
5. Chronic widespread pain or somatoform disorder (e.g. fibromyalgia).
6. Prior cervical medial branch radiofrequency neurotomy.
7. Severe clinical depression or psychotic features.
8. Possible pregnancy or other reason that precludes the use of fluoroscopy.
9. Daily chronic opiate use of >50 morphine equivalents.
10. Presence of pacemaker of neurostimulator.
11. Systemic infection at time of procedure.
12. Uncontrolled bleeding diathesis.
13. Requirement of IV procedural sedation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Post Procedure Pain Response | 3, 6, and 12 months
  Proportion of patients with a successful pain response (defined as ≥50% improvement in index pain) to Trident (T-CMBRFA) versus conventional (C-CMBRFA)

SECONDARY OUTCOMES:
Post Procedure Disability Response | 3, 6, and 12 months
  The proportion of patients with a successful functional response (defined as ≥ 10% reduction on neck disability index [NDI]) to T-CMBRFA versus C-CMBRFA
Post Procedure Patient Impression of Change | 3, 6, and 12 months
  The proportion of patients with a successful perception of improvement (defined as a score ≥6 on the Patient Global Impression of Change [PGIC]) to T-CMBRFA versus C-CMBRFA
Procedural Radiation Dose | After procedure
  Differences in procedural patient radiation dose during T-CMBRFA versus C-CMBRFA.
Procedure discomfort | After procedure
  Differences in procedural patient discomfort during T-CMBRFA versus C-CMBRFA.
Procedure time | After procedure
  Differences in procedural time during T-CMBRFA versus C-CMBRFA.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Utah Farmington Health Center, Farmington, Utah
  - University of Utah Orthopaedic Center, Salt Lake City, Utah
  - University of Utah South Jordan Health Center, South Jordan, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lord SM, Barnsley L, Wallis BJ, McDonald GJ, Bogduk N. Percutaneous radio-frequency neurotomy for chronic cervical zygapophyseal-joint pain. N Engl J Med. 1996 Dec 5;335(23):1721-6. doi: 10.1056/NEJM199612053352302. PMID 8929263
- [Background] Barnsley L. Percutaneous radiofrequency neurotomy for chronic neck pain: outcomes in a series of consecutive patients. Pain Med. 2005 Jul-Aug;6(4):282-6. doi: 10.1111/j.1526-4637.2005.00047.x. PMID 16083457
- [Background] McDonald GJ, Lord SM, Bogduk N. Long-term follow-up of patients treated with cervical radiofrequency neurotomy for chronic neck pain. Neurosurgery. 1999 Jul;45(1):61-7; discussion 67-8. doi: 10.1097/00006123-199907000-00015. PMID 10414567
- [Background] Cosman ER Jr, Dolensky JR, Hoffman RA. Factors that affect radiofrequency heat lesion size. Pain Med. 2014 Dec;15(12):2020-36. doi: 10.1111/pme.12566. Epub 2014 Oct 14. PMID 25312825
- [Background] Bogduk N E. International Spine Intervention Society. Cervical medial branch thermal radiofrequency neurotomy. Practice Guidelines: Spinal Diagnostic and Treatment Procedures, 2nd edition. 2013. 165-217 p.
- [Background] Finlayson RJ, Thonnagith A, Elgueta MF, Perez J, Etheridge JB, Tran DQ. Ultrasound-Guided Cervical Medial Branch Radiofrequency Neurotomy: Can Multitined Deployment Cannulae Be the Solution? Reg Anesth Pain Med. 2017 Jan/Feb;42(1):45-51. doi: 10.1097/AAP.0000000000000506. PMID 27776095
- [Background] Ebraheim NA, Haman ST, Xu R, Yeasting RA. The anatomic location of the dorsal ramus of the cervical nerve and its relation to the superior articular process of the lateral mass. Spine (Phila Pa 1976). 1998 Sep 15;23(18):1968-71. doi: 10.1097/00007632-199809150-00009. PMID 9779529
- [Background] Cohen SP, Strassels SA, Kurihara C, Lesnick IK, Hanling SR, Griffith SR, Buckenmaier CC 3rd, Nguyen C. Does sensory stimulation threshold affect lumbar facet radiofrequency denervation outcomes? A prospective clinical correlational study. Anesth Analg. 2011 Nov;113(5):1233-41. doi: 10.1213/ANE.0b013e31822dd379. Epub 2011 Sep 14. PMID 21918166
- [Background] Bogduk N. The clinical anatomy of the cervical dorsal rami. Spine (Phila Pa 1976). 1982 Jul-Aug;7(4):319-30. doi: 10.1097/00007632-198207000-00001. PMID 7135065
- [Background] Bogduk N, Kennedy DJ, Vorobeychik Y, Engel A. Guidelines for Composing and Assessing a Paper on Treatment of Pain. Pain Med. 2017 Nov 1;18(11):2096-2104. doi: 10.1093/pm/pnx121. PMID 28633460
- [Background] Pool JJ, Ostelo RW, Hoving JL, Bouter LM, de Vet HC. Minimal clinically important change of the Neck Disability Index and the Numerical Rating Scale for patients with neck pain. Spine (Phila Pa 1976). 2007 Dec 15;32(26):3047-51. doi: 10.1097/BRS.0b013e31815cf75b. PMID 18091500
- [Background] Harden RN, Weinland SR, Remble TA, Houle TT, Colio S, Steedman S, Kee WG; American Pain Society Physicians. Medication Quantification Scale Version III: update in medication classes and revised detriment weights by survey of American Pain Society Physicians. J Pain. 2005 Jun;6(6):364-71. doi: 10.1016/j.jpain.2005.01.350. PMID 15943958
- [Background] Ayearst L, Harsanyi Z, Michalko KJ. The Pain and Sleep Questionnaire three-item index (PSQ-3): a reliable and valid measure of the impact of pain on sleep in chronic nonmalignant pain of various etiologies. Pain Res Manag. 2012 Jul-Aug;17(4):281-90. doi: 10.1155/2012/635967. PMID 22891194
- [Background] Luedtke K, Basener A, Bedei S, Castien R, Chaibi A, Falla D, Fernandez-de-Las-Penas C, Gustafsson M, Hall T, Jull G, Kropp P, Madsen BK, Schaefer B, Seng E, Steen C, Tuchin P, von Piekartz H, Wollesen B. Outcome measures for assessing the effectiveness of non-pharmacological interventions in frequent episodic or chronic migraine: a Delphi study. BMJ Open. 2020 Feb 12;10(2):e029855. doi: 10.1136/bmjopen-2019-029855. PMID 32051295
- [Background] Walker E, Nowacki AS. Understanding equivalence and noninferiority testing. J Gen Intern Med. 2011 Feb;26(2):192-6. doi: 10.1007/s11606-010-1513-8. Epub 2010 Sep 21. PMID 20857339
- [Background] Kovacs FM, Abraira V, Royuela A, Corcoll J, Alegre L, Tomas M, Mir MA, Cano A, Muriel A, Zamora J, Del Real MT, Gestoso M, Mufraggi N; Spanish Back Pain Research Network. Minimum detectable and minimal clinically important changes for pain in patients with nonspecific neck pain. BMC Musculoskelet Disord. 2008 Apr 10;9:43. doi: 10.1186/1471-2474-9-43. PMID 18402665
- [Background] Julious SA. Sample sizes for clinical trials with normal data. Stat Med. 2004 Jun 30;23(12):1921-86. doi: 10.1002/sim.1783. PMID 15195324
- [Background] Chow JTY, Turkstra TP, Yim E, Jones PM. Sample size calculations for randomized clinical trials published in anesthesiology journals: a comparison of 2010 versus 2016. Can J Anaesth. 2018 Jun;65(6):611-618. doi: 10.1007/s12630-018-1109-z. Epub 2018 Mar 22. PMID 29569142
- See also: The burden of musculoskeletal diseases in the United States. — https://linkinghub.elsevier.com/retrieve/pii/S0049017216301445
- See also: The Prevalence of Cervical Zygapophyseal Joint Pain; A First Approximation. — http://journals.lww.com/00007632-199207000-00003
- See also: The Prevalence of Chronic Cervical Zygapophysial Joint Pain After Whiplash. — http://journals.lww.com/00007632-199501000-00004
- See also: False-Positive Rates of Cervical Zygapophysial Joint Blocks. — http://journals.lww.com/00002508-199306000-00007
- See also: Medial branch blocks are specific for the diagnosis of cervical zygapophyseal joint pain. — http://www.ncbi.nlm.nih.gov/pubmed/8117629
- See also: Radiofrequency neurotomy for the treatment of third occipital headache. — https://jnnp.bmj.com/lookup/doi/10.1136/jnnp.74.1.88
- See also: Core outcome measures for chronic pain clinical trials: IMMPACT recommendations. — http://content.wkhealth.com/linkback/openurl?sid=WKPTLP:landingpage&an=00006396-200501000-00005
- See also: Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. — https://journals.lww.com/00006396-200111000-00006